CLINICAL TRIAL: NCT00118066
Title: A Randomized Phase II Trial Of Calcitriol In Patients With Prostatic Intraepithelial Neoplasia
Brief Title: Calcitriol in Preventing Prostate Cancer in Patients With Prostatic Intraepithelial Neoplasia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accruaL, lack of scientific progress
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Rutgers Cancer Institute of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 080404; P30CA072720 (NIH); CDR0000433508 (Other: NIH); 0220044901 (Other: CINJ IRB); CINJ-NJ3803
Record Dates: First submitted 2005-07-08; First posted 2005-07-11 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Precancerous/Nonmalignant Condition; Prostate Cancer
Keywords: prostate cancer; high grade prostatic intraepithelial neoplasia
MeSH Terms: conditions — Precancerous Conditions; Prostatic Neoplasms | interventions — Calcitriol; Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Experimental): Patients receive oral calcitriol once daily for 8 weeks. Treatment repeats every 8 weeks for 2 courses. After completion of course 2 (week 16), patients undergo biopsy. Patients continue to receive calcitriol for up to 3 additional weeks while the biopsy is being evaluated. Patients with persistent high-grade prostatic intraepithelial neoplasia (HGPIN) by biopsy receive 2 additional courses of calcitriol.
  Interventions: Dietary Supplement: calcitriol
- Arm II (Other): Patients undergo observation for 16 weeks. At week 16, patients undergo biopsy. Patients with persistent HGPIN by biopsy receive 2 courses of calcitriol as in arm I.
  Interventions: Dietary Supplement: calcitriol; Procedure: observation

INTERVENTIONS:
Dietary Supplement: calcitriol — Given orally
Procedure: observation — No initial intervention
  Arms: Arm II

SUMMARY:
RATIONALE: Chemoprevention is the use of certain drugs to keep cancer from forming, growing, or coming back. The use of calcitriol may prevent prostate cancer. It is not yet known whether calcitriol is more effective than observation in preventing prostate cancer.

PURPOSE: This randomized phase II trial is studying how well calcitriol works in preventing prostate cancer in patients with prostatic intraepithelial neoplasia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the effects of calcitriol in patients with high-grade prostatic intraepithelial neoplasia.
* Determine the toxicity of this drug in these patients.
* Determine the effect of this drug on prostate specific antigen in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 arms.

* Arm I: Patients receive oral calcitriol once daily for 8 weeks. Treatment repeats every 8 weeks for 2 courses in the absence of unacceptable toxicity.

After completion of course 2 (week 16), patients undergo biopsy. Patients continue to receive calcitriol for up to 3 additional weeks while the biopsy is being evaluated. Patients with persistent high-grade prostatic intraepithelial neoplasia (HGPIN) by biopsy receive 2 additional courses of calcitriol. Patients with no HGPIN or prostate cancer by biopsy are removed from the study.

* Arm II: Patients undergo observation for 16 weeks. At week 16, patients undergo biopsy. Patients with persistent HGPIN by biopsy receive 2 courses of calcitriol as in arm I. Patients with no HGPIN or prostate cancer by biopsy are removed from the study.

After completion of study treatment, patients are followed annually for 2 years.

PROJECTED ACCRUAL: A total of 50 patients (25 per arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed high-grade prostatic intraepithelial neoplasia

  * Diagnosed within the past 6 months
* No evidence of prostate cancer within the past 6 months
* No evidence of palpable nodules on digital rectal exam
* Prostate specific antigen ≤ 10 ng/mL within the past 3 months

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* SGOT and SGPT ≤ 1.5 times upper limit of normal

Renal

* No uncontrolled renal failure
* No cancer-related hypercalcemia or kidney stones within the past 5 years

Cardiovascular

* No uncontrolled coronary artery disease
* No uncontrolled congestive heart failure

Other

* Prior malignancy allowed provided patient was curatively treated and has been disease-free for an appropriate time period for the specific cancer
* No known HIV positivity
* No active infection
* No major depression or suicidal ideation
* No other condition that would preclude study compliance
* No other uncontrolled medical condition

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy for any malignancy

Endocrine therapy

* At least 2 weeks since prior and no concurrent finasteride (Prosear® or Propecia®) or other androgen suppressor
* No concurrent corticosteroids

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* At least 2 weeks since prior phenytoin or phenobarbital
* At least 2 weeks since prior ketoconazole
* No concurrent administration of any of the following:

  * Magnesium-containing antacids
  * Thiazide diuretics
  * Calcium supplements
  * Digoxin
  * Herbal supplements
  * Pharmacological doses of cholecalciferol (vitamin D) or its derivatives

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2004-05; Primary Completion 2011-06 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Presence of prostate intraepithelial neoplasia after 16 weeks | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert S. DiPaola, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (5):
- United States (5):
  - Central Jersey Oncology Center, PA - East Brunswick, East Brunswick, New Jersey
  - Carol G. Simon Cancer Center at Morristown Memorial Hospital, Morristown, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Overlook Hospital, Summit, New Jersey